CLINICAL TRIAL: NCT03962582
Title: Clinical Evidence for Supported Spinal Curves in Wheelchair Seating: A Randomized Comparison
Brief Title: Supportive Wheelchair Back Compared to Fabric Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Craig Hospital (Other); Motion Concepts (Unknown); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Jessica Pedersen, Research Scientist, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00205806
Record Dates: First submitted 2019-04-22; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: comparing two different back support to access if there are postural and functional differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Supportive Back Comparison (Experimental): Motion Concepts matrx back to be attached to individual's wheelchair in place of the individual's back. It will be adjusted for size and to support the spinal curves as compared to a fabric back
  Interventions: Device: Matrix back

INTERVENTIONS:
Device: Matrix back — The Matrix back will replace the individual's back and the measures will be taken.

SUMMARY:
This study tests using a wheelchair back that supports the spine in a neutral position and one that allows the spine and pelvis to fall into a posterior pelvic tilt.

DETAILED DESCRIPTION:
Individuals will randomly start with the supportive back vs the unsupportive back. Measurements of the spine and pelvis will be taken. Forward upward reach, one stroke push, times forward push and ramp skills will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* complete spinal cord injury with levels
* Full time wheelchair users
* English speaking in order to understand the consent

Exclusion Criteria:

* Over 250 pounds in body weight
* Inability to grip a wheelchair push rim
* Individual with pressure ulcer
* Individual with shoulder pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Seated Body Measurements performed. | 2 hour session (one visit)
  Angle measurements will be taken when sitting. These include the pelvic angle (femur to pelvis) and Spinal Angle of Kyphosis (femur to acromion).
Vertical Forward Reach Test (VFRT): | 2 hour session (one visit)
  Assesses stability by measuring the maximum distance an individual can reach forward vertically (upward) while sitting in a fixed position.
Breathing status: | 2 hour session (one visit)
  An instrument called a spirometer is placed into the mouth with the nose clipped and the individual is instructed to take a deep breath and blow out. Peak effort flow, peak cough flow, and functional capacity will be recorded.
One stroke push: | 2 hour session (one visit)
  This measures how far the wheelchair moves forward with one stroke over carpet.
Timed forward Wheeling/Wheelchair Propulsion Test (WPT): | 2 hour session (one visit)
  The WPT is a brief test measuring the number of wheelchair pushes and time needed to cross a distance of 23 meters
Ramp Ascent (forward wheeling | 2 hour session (one visit)
  This is a timed test on a 10.3 meter ramp with a 1:13 grade slope
Pain Scale: | 2 hour session (one visit)
  The participant will rate any pain felt while sitting in the test wheelchairs after all activities using a numerical scale of 0-10, with 0 being no pain.
Survey | 2 hour session (one visit)
  The study team developed a survey for patients to fill out asking questions such as comfort of back support and opinions of practicality of back support.

SECONDARY OUTCOMES:
Breathing status: | 2 hour session (one visit)
  Pulse oximetry will be taken with the person sitting in each testing wheelchair.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No